CLINICAL TRIAL: NCT01058993
Title: A Phase I Study of the CXCR-4 Inhibitor AMD3100 for the Treatment of Neutropenia Due to Mutations of CXCR-4, the Myelokathexis Syndrome
Brief Title: AMD 3100 for Treatment of Myelokathexis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, David Dale, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35419-D; MAMO-0407-1 (Other: Protocol ID #)
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Results first posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-05

CONDITIONS: Neutropenia
Keywords: neutropenia; myelokathexis; WHIM syndrome; AMD 3100; plerixafor; Myelokathexis syndrome; Neutropenia due to mutations of CXCR-4
MeSH Terms: conditions — Neutropenia; WHIM syndrome | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMD3100 or plerixafor (Experimental): SINGLE arm study with increasing doses of Plerixafor
  Interventions: Drug: AMD3100 or plerixafor

INTERVENTIONS:
Drug: AMD3100 or plerixafor — The study will examine the hematological effects/safety of plerixafor in patients with myelokathexis attributable to mutations of CXCR4. Plerixafor will be administered on days 1, 3, 5, 8, and 10. Five intrapatient escalating doses of AMD 3100, 20 micrograms per kilogram (mcg/kg), 40 micrograms per kilogram (mcg/kg), 80 micrograms per kilogram (mcg/kg), and 240 micrograms per kilogram (mcg/kg) will be examined in the patients at University of Washington General Clinical Research Center for up to 10 days, requiring subjects be available up to 14 days. Patients will be monitored for hematological effects of plerixafor and observed for adverse effects. If normal blood neutrophil count is achieved and maintained for at least 24 hours prior to highest dose, we will stop at that level.
  Other Names: Mozobil

SUMMARY:
This is an initial study to determine if CXCR4 inhibitor AMD 3100 or plerixafor may be a potential treatment for neutropenia due to CXCR4 mutations, the myelokathexis or WHIM (warts, hypogammaglobulinemia, immunodeficiency and myelokathexis) syndrome. This is the initial study of this concept and will involve up to 6 patients to receive increasing doses of plerixafor administered subcutaneously or on an alternate day basis. It is unknown if these patients will be highly sensitive to a blockade of CXCR4 activity and release more white blood cells than normal volunteers or cancer patients given the same dose of this drug. Therefore doses will begin at a level 12 fold less than currently used to mobilize stem cells and will be increased stepwise to achieve an acceptable circulating level of neutrophils.

DETAILED DESCRIPTION:
This is an open label, single Center, phase I study to examine the hematological effects, pharmacokinetics and safety of plerixafor in patients with myelokathexis attributable to mutations of CXCR4, utilizing serial, escalating doses of plerixafor administered on days 1, 3, 5, 8, and 10. Five intrapatient escalating dose levels, 20 micrograms per kilogram (mcg/kg), 40 micrograms/kilogram(mcg/kg), 80 micrograms/kilogram(mcg/kg), and 240 micrograms/kilogram (mcg/kg)will be examined. The subjects will be patients at the University of Washington General Clinical Research Center for up to 10 days; the study requires subject be available for up to 14 days. Patients will be monitored for hematological effects of plerixafor and observed for adverse effects. If a normal blood neutrophil count is achieved and maintained for at least 24 hours prior to the highest dose, we will stop at that level.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years, WBC (white blood count) less than 3.0 x 10^9 per Liter,
* Absolute neutrophil count less than 2.0 x 10^9 per Liter,
* platelets greater than 100 x 10^6 per Liter, creatinine less than 2.0/milligrams per/deciliter,
* Creatinine clearance > 60 ml/min calculated,
* Aspartate Aminotransferase-GOT (SGOT), Alanin Aminotransferase-GPT (SGPT), bilirubin < 2.5 upper limit of normal,
* Eastern Cooperative Oncology Group (ECOG) status 0 or 1,
* mutation identified and confirmed in CXCR4,
* on no granulocyte-colony stimulating factor (G-CSF), granulocyte-macrophage-colony stimulating factor (GM-CSF) within 3 weeks of the study drug
* patient signs consent, accepts contraception

Exclusion Criteria:

* greater than 18 years of age,
* sensitivity to plerixafor,
* pregnant,
* prisoner,
* decisionally impaired,
* judged unlikely to comply,
* illness that may interfere with interpretation of results,
* leukemia,
* malignancy,
* active infection requiring antibiotics within one week of study drug administration,
* history of cardiac conduction or electrocardiogram (EKG) abnormality,
* previous experimental therapy within one week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Dale, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Dale DC, Bolyard AA, Kelley ML, Westrup EC, Makaryan V, Aprikyan A, Wood B, Hsu FJ. The CXCR4 antagonist plerixafor is a potential therapy for myelokathexis, WHIM syndrome. Blood. 2011 Nov 3;118(18):4963-6. doi: 10.1182/blood-2011-06-360586. Epub 2011 Aug 11. PMID 21835955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were contacted from the Severe Chronic Neutropenia International Registry office by Audrey Anna Bolyard, Manager of the Registry.
Pre-assignment Details: Prior to assignment, we performed physician, EKG (electrocardiogram) and screening labs, including CBC (complete blood count), Differential and smear, comprehensive metabolic panel, urinalysis, and pregnancy testing on females subjects
Groups:
- Single Arm Study, 5 Escalating Doses of AMD3100 (Plerixafor): Single arm study to examine the hematological effects, pharmacokinetics and safety of plerixafor in patients with myelokathexis attributable to mutations of CXCR4, utilizing serial, escalating doses of plerixafor administered on days 1, 3, 5, 8, and 10. Five intrapatient escalating dose levels, 20 micrograms per kilogram (mcg/kg), 40 micrograms/kilogram(mcg/kg), 80 micrograms/kilogram(mcg/kg), and 240 micrograms/kilogram (mcg/kg)will be examined. The subjects will be patients at the University of Washington General Clinical Research Center for up to 10 days; the study requires subject be available for up to 14 days. Patients will be monitored for hematological effects of plerixafor and observed for adverse effects. If a normal blood neutrophil count is achieved and maintained for at least 24 hours prior to the highest dose, we will stop at that level.
Period: Overall Study
Arm/Group | Single Arm Study, 5 Escalating Doses of AMD3100 (Plerixafor)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study, 5 Escalating Doses of AMD3100 (Plerixafor)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.7 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6
Blood neutrophil count (in myelokathexis) [Mean (Full Range); unit: 10^9 per Liter] | 0.7 [0.2 to 1.8]
blood neutrophil levels [Mean (Standard Deviation); unit: 10^9 per Liter] — On days 1, 3, 5, 8 and 10 a small sample of blood was drawn for CBC, Differential and Smear Evaluation, performed for determination of blood cell counts before and at 30 minutes, 1, 2, 4, 6, 9 and 12 hours after the drug was given. This required placement of a catheter that was left in place for 12 hours for ease of serial blood sampling. On the days between injections of plerixafor/AMD3100, a sample of blood was taken once in the morning via a needle in an arm vein.
  10^9 per Liter | 0.7 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Blood Neutrophil Counts.
Description: Effectiveness of drug based on increases of blood neutrophil counts to greater than 2.0 x 10^9 per liter
Time Frame: up to 14 days, depending on when subject reached peak response, i.e., the highest count after the stimulus (plerixafor)
Population: The number of participants (6) was determined by the fact that we were studying a rare form of neutropenia, WHIMS syndrome, and we therefore recruited subjects who have WHIMS who live on the West coast. Analysis was per protocol.
Measure: Mean (Standard Deviation); unit: 10^9 per Liter
Arm/Group | SINGLE Arm Study, 5 Escalating Doses of AMD3100 (Plerixafor)
Number analyzed (Participants) | 6
10^9 per Liter | 4.48 (1.91)
Statistical Analysis 1: Comparison: SINGLE Arm Study, 5 Escalating Doses of AMD3100 (Plerixafor); Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Student t-test-comparison means of normal subjects & controls
Statistical Analysis 2: Comparison: SINGLE Arm Study, 5 Escalating Doses of AMD3100 (Plerixafor); The patients' leukocyte counts before and after plerixafor were compared; Test type: Superiority or Other; p < 0.05, Ratio paired t-test; Ratio paired t-test for comparison of baselines and responses for each category of leukocytes

ADVERSE EVENTS:
Arm/Group | Single Arm Study, 5 Escalating Doses of AMD3100 (Plerixafor)
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No